CLINICAL TRIAL: NCT00206141
Title: Multi-centre, Double-blind, Randomised, Parallel-group, Placebo-controlled, Phase 3 Study of the Efficacy & Safety of Quetiapine Fumarate & Lithium as Monotherapy in Adult Patients With Bipolar Depression for 8 Weeks & Quetiapine in Continuation (Abbreviated)
Brief Title: Seroquel in Bipolar Depression Versus Lithium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1447C00001; EMBOLDEN I
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Bipolar Disorder; Bipolar Depression; Depression
Keywords: Bipolar disorder; bipolar depression; depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Quetiapine Fumarate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Quetiapine Fumarate (Seroquel™) drug, mood stabilizer (mood)

SUMMARY:
This study is being carried out to see if quetiapine fumarate (Seroquel) is effective in treating bipolar depression during an 8-week acute phase compared with placebo and lithium, followed by continuation treatment for 26 up to 52 with quetiapine fumarate (Seroquel) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of bipolar I disorder or bipolar II disorder, currently depressed, aged 18 to 65 years old and outpatient status at enrolment and randomization.

Exclusion Criteria:

* Patients with a current DSM-IV Axis I disorder other than bipolar disorder that is symptomatic or requiring treatment within 6 months of enrolment,
* History of non-response to an adequate treatment
* Patients who, in the investigator's judgment pose a current serious suicidal or homicidal risk
* Pregnancy or lactation
* Clinically relevant disease or clinical finding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672
Dates: Start 2005-08; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The change from randomization to Week 8 assessment in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score.

SECONDARY OUTCOMES:
MADRS total score response
MADRS total score remission

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (76):
- Canada (9):
  - Research Site, Kelowna, British Columbia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
- Croatia (4):
  - Research Site, Osijek
  - Research Site, Split
  - Research Site, Zadar
  - Research Site, Zagreb-Susedgrad
- Estonia (3):
  - Research Site, Kohtla-Järve
  - Research Site, Tallinn
  - Research Site, Tartu
- Germany (2):
  - Research Site, Berlin
  - Research Site, Würzburg
- Indonesia (3):
  - Research Site, Solo, Java
  - Research Site, Jakarta
  - Research Site, Lawang
- Latvia (2):
  - Research Site, Daugavpils
  - Research Site, Riga
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Šiauliai
  - Research Site, Vilnius
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching Sarawak
  - Research Site, Petaling Jaya
- Norway (5):
  - Research Site, Brattvåg
  - Research Site, Drammen
  - Research Site, Fredrikstad
  - Research Site, Mysen
  - Research Site, Paradis
- Philippines (4):
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Mandaluyong
  - Research Site, Manila
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdynia
  - Research Site, Leszno
  - Research Site, Lodz
  - Research Site, Skorzewo
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Russia (12):
  - Research Site, Arkhangelsk
  - Research Site, Kazan'
  - Research Site, Lipetsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Stavropol
  - Research Site, Tver'
  - Research Site, Yaroslavl
- Serbia (5):
  - Research Site, Belgrade
  - Research Site, Čačak
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Valjevo
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Taiwan (2):
  - Research Site, Changhua
  - Research Site, Taipei
- Ukraine (9):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Luhansk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Simferopol
  - Research Site, Vinnitsa

REFERENCES:
- [Derived] Young AH, McElroy SL, Bauer M, Philips N, Chang W, Olausson B, Paulsson B, Brecher M; EMBOLDEN I (Trial 001) Investigators. A double-blind, placebo-controlled study of quetiapine and lithium monotherapy in adults in the acute phase of bipolar depression (EMBOLDEN I). J Clin Psychiatry. 2010 Feb;71(2):150-62. doi: 10.4088/JCP.08m04995gre. Epub 2010 Jan 26. PMID 20122369